CLINICAL TRIAL: NCT04163146
Title: Lung Function Variability in Children and Adolescents
Acronym: LUV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Patras (Other)
Responsible Party: Principal Investigator, Fouzas Sotirios, Assistant Professor of Pediatrics, University of Patras
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LUV_2019
Record Dates: First submitted 2019-11-09; First posted 2019-11-14 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Asthma in Children; Lung Function Decreased
Keywords: Asthma; Lung function variability; Children; Adolescents
MeSH Terms: conditions — Respiratory Insufficiency; Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy children and adolescents (Experimental): Healthy children and adolescents aged 6 to 18 years (N=100) for the assessment of normal PEF and FEV1 variability.
  Interventions: Diagnostic Test: Measurements of PEF and FEV1
- Asthmatic children and adolescents (Experimental): Children and adolescents aged 6 to 18 years with diagnosed asthma (N=100) for the assessment of PEF and FEV1 variability in asthmatics.
  Interventions: Diagnostic Test: Measurements of PEF and FEV1

INTERVENTIONS:
Diagnostic Test: Measurements of PEF and FEV1 — Measurements of PEF and FEV1 at home, twice a day (07:00 - 09:00 and 19:00 - 21:00) and for a period of 3 months, using portable spirometers connected to smartphone

SUMMARY:
Long-term variability analysis of peak expiratory flow (PEF) and forced expiratory volume in 1 s (FEV1) has been successfully used in research to predict the exacerbation of the disease in adult individuals with asthma. However, there is a paucity of data regarding PEF and FEV1 variability in asthmatic children and adolescents. Such a task requires at least daily PEF and FEV1 measurements, recording in diaries, and periodic evaluation of the data. The process may be proven both complicated and time consuming, thus reducing patients' adherence. Recent advances in biosensor technology have permitted the development of reliable, low-cost, portable spirometers, able to connect with smartphones and monitor lung function parameters in real time and from a distance.

The objectives of the present study is the assessment of PEF and FEV1 variability: a) in healthy children and adolescents, in order to define the normal daily fluctuation of PEF and FEV1 and the parameters that may influence it, and b) in children and adolescents with asthma, in order to explore the differences from healthy subjects and reveal any specific variability changes prior to exacerbation. Such data would improve our understanding regarding the disease and permit the development of integrated tools for assessing the level of asthma control and the risk of future exacerbations.

The study will include 100 healthy children and adolescents aged 6 to 18 years for the assessment of normal PEF and FEV1 variability, and 100 children and adolescents of the same age with diagnosed asthma for the assessment of PEF and FEV1 variability in asthmatics. PEF and FEV1 measurements will be performed using an FDA-approved portable spirometer (MIR Spirobank Smart) capable to connect to smartphone. Each participant will receive his personal spirometer. Measurements will be performed twice a day between 07:00-09:00 and 19:00-21:00 hours and dispatched via email to a central database for a period of 3 months. PEF and FEV1 variability will be assessed by detrended fluctuation analysis, aiming to define the normal pattern (healthy controls) and to detect and quantify the deviations (asthmatics). The anticipated duration of the study is 24 months.

DETAILED DESCRIPTION:
Background

Asthma represents the most common chronic disease of childhood and adolescence and an important cause of morbidity worldwide. The disease is characterized by episodes of reversible airway obstruction (exacerbations), associated with specific symptoms (wheeze, dyspnea, cough, chest tightness) and decrease in peak expiratory flow (PEF) and forced expiratory volume at 1 sec (FEV1). However, these spirometric changes occur in parallel with clinical deterioration, thus presenting limited ability to predict the exacerbation of the disease.

Both PEF and FEV1 demonstrate significant daily variability, i.e., circadian and/or day-by-day fluctuation of the measured values. In healthy individuals the pattern of these fluctuations remains constant over long time periods (weeks, months), as opposed to asthmatic patients where PEF and FEV1 variability is increased, especially prior to exacerbations when the control of the disease is lost. Thus, the analysis of PEF and FEV1 variability has been used in research to evaluate the effectiveness of treatment, recognize high-risk patients and predict asthma exacerbations.

In clinical practice, however, the evaluation of PEF and FEV1 variability requires at least daily measurements with special devices, recording in diaries, and periodic evaluation of the data by the attending physicians. The process may be proven both complicated and time consuming, thus reducing patients' adherence especially in the case of asthmatic children and adolescents. In addition, the periodic review of measurements may hamper the prediction of exacerbation, as the time of evaluation may not coincide with changes in the variability of lung function that characterize the loss of asthma control.

Over the last years, technological advancements in the field of biosensors and microprocessors have permitted the development of reliable, low-cost, portable spirometers, able to connect with cutting-edge mobile phones (smartphones) and monitor lung function parameters in real time and from a distance. The use of such devices may overcome most of the aforementioned barriers in following-up lung function parameters in the long term.

Currently, there is a paucity of data regarding PEF and FEV1 variability in children and adolescents with asthma. Such data would improve our understanding regarding the disease and permit the development of integrated tools for assessing the level of asthma control and the risk of future exacerbations

Objectives

The objectives of the study are:

1. Assessment of PEF and FEV1 variability in healthy children and adolescents: definition of the normal range of daily PEF and FEV1 fluctuation and the parameters that may influence it
2. Assessment of PEF and FEV1 variability in children and adolescents with asthma: differences from healthy subjects and definition of specific changes prior to exacerbation

   Methods

   A. Study population

   The study will include two cohorts:
   1. Healthy children and adolescents aged 6 to 18 years (N=100) for the assessment of normal PEF and FEV1 variability (objective #1).
   2. Children and adolescents aged 6 to 18 years with diagnosed asthma [2] (N=100) for the assessment of PEF and FEV1 variability in asthmatics (objective #2).

   B. Lung function measurements

   a. Device: PEF and FEV1 measurements will be performed using an FDA-approved portable spirometer (Spirobank Smart, MIR, Rome, Italy), with a disposable bi-directional digital turbine (flow range ±16L/s, volume accuracy ±3% or 50 mL, flow accuracy: ±5% or 200 mL/s, dynamic resistance <0.5 cm H2O/L/s), capable to connect to smartphone via Bluetooth® using a dedicated freeware application (iSpirometry, MIR, Rome, Italy). Each participant will receive his personal spirometer. Detailed information regarding the use and maintenance of the device will be provided (brochure & online resources).

   b. Measurements: The correct technique for PEF and FEV1 measurements (ERS/ATS standards) will be demonstrated by one of the investigators at enrollment. Detailed information regarding the technique (brochure & online resources) will be also provided. Measurements will be performed twice a day between 07:00-09:00 and 19:00-21:00 hours, for a period of 3 months.

   c. Completed measurements (encrypted pdf format) will be dispatched via email to a central database by the participants or their parents.

   d. Monitoring: Participants' adherence will be monitored continuously. The investigators will notify the participants in case of lost measurements or inappropriate technique.

   C. Variability analysis

   PEF and FEV1 variability will be assessed by:

   a. The coefficient of variation b. Detrended Fluctuation Analysis (DFA), a method that has been widely used for the investigation of intrinsic correlation within time series.14 Initially, the square root of the time series [F(n)] is calculated for segments of different (time) length n. A linear relationship in the logarithmic graph F (n) - log (n) indicates the existence of fractal architecture in the scaling of the specific data, while the slope a of the line describes the pattern of long-term fluctuations.14 A change in daily variability of PEF or FEV1 results in a simultaneous deviation from the predetermined a value.6 This deviation can easily be detected and quantified. It has been shown that the magnitude of a deviation reflects the likelihood of asthma exacerbation within the next month.6 c. Variability analysis will be performed in MatLab (MathWorks, Inc., Natick, MA, USA) environment.

   D. Additional data Patients' characteristics (age, sex, baseline lung function, allergy, comorbidities, medication, etc) will be also recorded. These parameters will be included in regression models to explore their effect on the pattern of PEF and FEV1 variability.

   E. Statistics All analyses will be performed with the IBM SPSS software version 25.0 (IBM Corp., Armonk, NY).

   F. Timeframes The expected duration of the study is 24 months. • Part I: Assessment of PEF and FEV1 variability in healthy children and adolescents Duration: 9 months (January - September 2020).

   PEF and FEV1 measurements from 100 participants (3 months each)

   • Part II: Assessment of PEF and FEV1 variability in asthmatic children and adolescents Duration: 15 months (October 2020 - December 2021). PEF and FEV1 measurements from 100 participants (3 months each)

   G. Ethics The study will comply to the regulations and standards of good medical practice. Participants will receive a unique study number and no personal data will be recorded. Measurements will be dispatched via email in encrypted pdf format. Informed written parental consent will be obtained prior to enrollment. Children aged >12 years will also provide a written consent. The study has been approved by the Ethics Committee of the University Hospital of Patras, Greece (decision # 329/02-04-2019).

ELIGIBILITY:
Cohort A. Healthy children and adolescents

Inclusion Criteria:

* Age 6 - 18 years
* No asthma or asthma medication in the last 2 years
* Normal baseline spirometry
* Smartphone possession (parents or participants) with ability of internet connection (Wi-Fi or mobile data)
* Informed written consent (parents, parents & children >12 years old)

Exclusion Criteria:

* Inability to perform 3 consecutive measurements within the 3-month period of observation
* Inability to perform 6 measurements in total (3.3% of the anticipated 180 measurements) within the 3-month period of observation
* Major respiratory events (e.g., asthma attack, severe respiratory infection, chest trauma) or other health-related events that may hamper the performance of lung function measurements (e.g., surgery, trauma) within the 3-month period of observation.

Cohort B. Children and adolescents with asthma

Inclusion Criteria:

* Age 6 - 18 years
* Doctor-diagnosed asthma under treatment
* Smartphone possession (parents or participants) with ability of internet connection (Wi-Fi or mobile data)
* Informed written consent (parents, parents & children >12 years old)

Exclusion Criteria:

* Inability to perform 3 consecutive measurements within the 3-month period of observation
* Inability to perform 6 measurements in total (3.3% of the anticipated 180 measurements) within the 3-month period of observation
* Major respiratory events (e.g., severe respiratory infection, chest trauma) or other health-related events that may hamper the performance of lung function measurements (e.g., surgery, trauma) within the 3-month period of observation

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
PEF variability | 3 months
  Daily fluctuations in PEF values
FEV1 variability | 3 months
  Daily fluctuations in FEV1 values

CONTACTS AND LOCATIONS:
Overall Officials: Sotirios Fouzas, Study Chair — University of Patras
Locations (1):
- Pediatric Respiratory Unit, University Hospital of Patras, Pátrai, Achaia, Greece

REFERENCES:
- [Derived] Frima ES, Theodorakopoulos I, Gidaris D, Karantaglis N, Chatziparasidis G, Plotas P, Anthracopoulos M, Fouzas S. Lung Function Variability in Children and Adolescents With and Without Asthma (LUV Study): Protocol for a Prospective, Nonrandomized, Clinical Trial. JMIR Res Protoc. 2020 Aug 7;9(8):e20350. doi: 10.2196/20350. PMID 32763874